CLINICAL TRIAL: NCT02676921
Title: Phase 1: Study of the Osteogenic Potential of Human Maxillary Sinus Shneiderian Membrane
Brief Title: The Osteogenic Potential of Human Maxillary Sinus Shneiderian Membrane
Acronym: HMSSM
Status: Completed | Type: Observational
Sponsor: BERBERI ANTOINE (Other)
Collaborators: Lebanese University (Other)
Responsible Party: Sponsor-Investigator, BERBERI ANTOINE, Professor, Lebanese University
Organization: Lebanese University (Other)
Other Study IDs: 18840
Record Dates: First submitted 2015-09-06; First posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Sinus; Empyema, Maxillary (Chronic)
Keywords: sinus membrane; osteogenic
MeSH Terms: conditions — Fistula; Empyema; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — Human sinus membrane
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- GROUP 1: Ten samples of sinus membrane where harvested from fifteen patients during a surgical nasal approach for treatment of chronic rhinosinusitis.

SUMMARY:
The objectives of this study are :

1. to test the the osteogenic potential of human maxillary sinus schneiderian membrane (hMSSM).
2. To investigate the expression of mesenchymal stem cell marker (STRO-1), a marker of mesenchymal progenitor cells using flow cytometry, and Alkaline phosphate expression, Red alizarin and Von Kossa staining and quantitive PCR.

DETAILED DESCRIPTION:
1. Isolation and Culture of hMSM-Derived Cells.

   The tissue will be washed again with Phosphate Buffered Saline (PBS) that included antibiotic and antimytotic, cut into small pieces under aseptic conditions, treated with 0.06% collagenase type II (In vitrogen) and dispase, shaken with an incubator (CO2 incubator, Forma Scientific) containing 5% CO2 at 37°C for 4 hours, and centrifuged at 1,000 (Revolution Per Minute) for 10 minutes (large-capacity tabletop centrifuge).
   * The precipitate was suspended in an alpha minimum essential medium (α-MEM) (Sigma-Aldrich) containing 10% fetal bovine serum and 1% penicillin-streptomycin and filtered with a 40-μm cell strainer (BD Bioscience), with which all tissues except for the hMSSM-derived cells were filtered out.
   * The solution filtered out was cultured in an incubator. Daily morphologic characteristics will be observed with an inverted microscope, and the culture solution will be changed every other day. When the medium will be changed, cells not adherent to the culture plate will be removed and only the adherent cells will be cultured. When the culture dishes become nearly confluent, the cells will be separated with Trypsin-ethylenediaminetetraacetic acid (EDTA) and subsequently repeated for continued passaging. The cells will be assayed at passage 3 for their osteogenic potential.
2. Flow Cytometry. Fluorescence-activated cell sorting (FACS) analysis for the expression of osteoprogenitor cell markers was performed on samples from primary cells (P0), passage 1 (P1) cultures, and passage 2 (P2) cultures cultured in nonosteogenic medium.

   Flow cytometry on the cell surface markers STRO-1, CD105, and CD146 for separation of Mesenchymal progenitor cells (MPCs) from hMSM will be conducted. The hMSSM-derived cells at passage 3 will be placed into a test tube (Becton- Dickinson) by 1 x104 cells/mL and washed three times with wash buffer (0.2% bovine serum albumin, 0.1% sodium azide, 0.5 mmol/L EDTA). The antibodies of CD146 (BD Bioscience) and CD105 (BD Bioscience) to which fluorescein isothiocyanate and phycoerythrin were adhered will be treated for 1 hour and washed with wash buffer three times, and the origin of stem cell was observed with flow cytometry (BD bioscience). For STRO-1 (human antimouse monoclonal antibody, immunoglobulin M subclass; R&D Systems), antibody was treated for 1 hour and washed three times with wash buffer, and the secondary antibody, to which fluorescein isothiocyanate was attached, was treated for 30 minutes, washed three times with wash buffer, and observed with flow cytometry.
3. Osteogenic Differentiation of hMSM

   The hMSM-derived cells at passage 3 were incubated in osteogenic media for 1 to 4 weeks in 12 well plates at a density of 105 cells per well and divided into two groups. The control group was replated in a normal medium (complete α-MEM), and the experimental group was replated in osteogenic differentiation medium (α-MEM including 0.1 μm dexamethasone, 10 μm glycerol phosphate, and 50 μm L-ascorbic acid 2-phosphate). The media were changed every 3 days.

   3.1- Alkaline Phosphatase and Alizarin Red Staining. Control and experimental cultures were each washed three times with sterile triple-distilled water at 7, 14, 21, and 28 days after the treatment date, fixed with citrate-acetone- formaldehyde fixation solution (Sigma), and washed again three times with sterile triple-distilled water. They were then stained with an alkaline dye mixture (nitrite, Fast Red Violet-alkaline, naphthol alkaline solution; Sigma), in the dark for 15 minutes at normal temperature, washed three times with sterile triple-distilled water, counterstained with hematoxylin (Sigma), washed again three times with sterile triple-distilled water, and observed with an inverted microscope.

   Alizarin Red Staining. Control and experimental group samples were each washed three times with sterile triple-distilled water at 7, 14, 21, and 28 days from the treatment date, fixed with 4% paraformaldehyde (Merck) for 15 minutes, stained while light was isolated for 30 minutes with 2% alizarin red solution (Sigma), washed again three times with sterile triple-distilled water, and the staining will be observed with an inverted microscope.

   3.2- Von Kossa Staining. Control and experimental cultures were washed three times with sterile triple-dis- tilled water, fixed with 4% paraformaldehyde (Merck) at a normal temperature for 15 minutes and washed again three times with sterile triple-distilled water. They were stained for 30 minutes while light was isolated with 1% silver nitrate (Merck) solution, washed three times with sterile triple-distilled water, left under ultraviolet light for 1 hour, counterstained with 0.1% eosin (Sigma), and the staining will be observed with an inverted microscope.

   3.3- Quantitative PCR (qPCR). To observe osteocalcin expression, the hMSM-derived cells, differentiated into two groups, were washed with (PBS) at 7, 14, 21, and 28 days after treatment in osteogenic differentiation medium and collected with a cell scraper. After the Ribonucleic acid (RNA) was separated with an RNA extraction kit, it underwent a reverse-transcription reaction with the separated RNA, osteocalcin, or bone sialoprotein, or dentin matrix protein 1 primers and probes, and reverse-transcriptase polymerase chain reaction premix (Applied Biosystems). The obtained data will be normalized using 18 Shake. The amplified products were analyzed using the deal-delta Computer Tomography analysis.
4. Histochemical staining of alkaline phosphatase activity in frozen sections of sinus mucosa.

   Freshly prepared sinus mucosa was washed in phosphate-buffered saline (PBS), cut into pieces of approximately 5x 5 mm, embedded in optimum cutting temperature tissue compound (OCT compound; Miles Laboratories, USA), and stored at - 80 C. Frozen sections (7 mm) mounted on poly-D-lysine-coated slides were fixed with ice-cold acetone for 1 min and allowed to air dry. The slides were washed with PBS and subsequently incubated with the substrate solution for alkaline phosphatase activity containing 4 mg of naphthol phosphate in 0.15 ml of N, N0 -dimethyl- formamide and 12mg of fast blue salt (Sigma, St Louis, USA) in 15 ml of Tris-Hydrogen Chloride (pH 9.6). After rinsing with distilled water, slides were counterstained with hematoxylin-eosin, embedded into water-soluble resin, and photographed.
5. Immunohistochemical determination of STRO-1-positive cells in frozen sections of mucosa.

Frozen sections (7 mm) were fixed with cold acetone for 1 min and washed in PBS. The slides were placed into PBS containing 0.3% of hydrogen peroxide for 15 minutes to quench endogenous peroxidase, washed, and blocked with 2% bovine serum albumin in PBS for 1hour at room temperature. Sections were incubated with a 1: 50 dilution of the STRO-1 antibody (mouse monoclonal antibody, IgM subclass; Developmental Studies Hybridoma Bank, University of Iowa, USA) in blocking solution overnight at 41 degree C. For detection of STRO-1-positive cells, slides were incubated with a biotinylated goat anti-mouse Immune globulin M (IgM) (1 : 100, An der Grub, Vienna, Austria) and a streptavidin-peroxidase conjugate (BioFX Laboratories, Inc., MD, USA) each at room temperature for 45 min. The peroxidase-containing complex was visualized by Diaminobenzidine substrate (Dako, Glostrup, Denmark) and counterstained with hematoxylin. The sections were embedded into water-soluble resin and photographed.

ELIGIBILITY:
Inclusion Criteria:

* Patients, (n = 10), who suffered from posterior or total maxillary excess undergoing posterior or total maxillary superiorly impaction for orthognathic surgery. These patients do not present any pathological issues in the maxillary sinus
* Patients, (n = 10), who suffered from a sinus problem and needs a surgical nasal approach. These patients have an inflammatory or an ongoing disease process in the maxillary sinus

Exclusion Criteria:

* Smokers or patients with skeletal disorders and syndromatic diseases will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The present study investigates whether human sinus Shneiderian membrane (hMSSM) contain an osteogenic progenitor cell population capable of forming bone by utilizing in vitro assays.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Isolation and Culture of hMSM-Derived Cells - Flow Cytometry | 3 months
  The tissue will be washed again with PBS that included antibiotic and antimycotic , cut into small pieces under aseptic conditions, treated with 0.06% collagenase type II and Dispase, shaken with an incubator containing 5% CO2 at 37°C for 4 hours, and centrifuged at 1,000 RPM for 10 minutes
  * The precipitate was suspended in an alpha minimum essential medium containing 10% fetal bovine serum (Hyclone) and 1% penicillin-streptomycin and filtered with a 40-μm cell strainer , with which all tissues except for the hMSM-derived cells were filtered out.
  * The solution filtered out was cultured in an incubator. Daily morphologic characteristics will be observed with an inverted microscope, and the culture solution will be changed every other day. When the medium will be changed, cells not adherent to the culture plate will

CONTACTS AND LOCATIONS:
Overall Officials: Antoine N BERBERI, Ph.D, Principal Investigator — DENTAL SCHOOL LEBANESE UNIVERSITY
Locations (1):
- PRASE, Beirut, Lebanon

REFERENCES:
- [Derived] Bou Assaf R, Zibara K, Fayyad-Kazan M, Al-Nemer F, Cordahi M, Khairallah S, Badran B, Berberi A. Healing of Bone Defects in Pig's Femur Using Mesenchymal Cells Originated from the Sinus Membrane with Different Scaffolds. Stem Cells Int. 2019 Sep 30;2019:4185942. doi: 10.1155/2019/4185942. eCollection 2019. PMID 31662765